CLINICAL TRIAL: NCT01788306
Title: A Trial to Prevent Opioid Overdose: E.D. Based Intervention & Take-home Naloxone
Brief Title: Project OOPEN: Opioid Overdose Prevention, Education and Intervention
Acronym: OOPEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Caleb Banta-Green, Research Scientist, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 43874; 1R01DA030351 (NIH)
Record Dates: First submitted 2013-02-01; First posted 2013-02-11 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Opioid Overdose
Keywords: Elevated risk; opioid overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (OOPEN+BBCC) (Active Comparator): Study intervention, overdose prevention, education, intervention, brief behavioral change counseling, take-home naloxone, referral to local available resources.
  Interventions: Drug: OOPEN+BBCC
- Control (No Intervention): Standard of care, referral to local available resources.

INTERVENTIONS:
Drug: OOPEN+BBCC — Take-home naloxone is offered as part of a behavioral prevention intervention to reduce the occurrence of future opioid overdose.
  Arms: Intervention (OOPEN+BBCC)

SUMMARY:
This prospective, randomized emergency department trial will study the effectiveness of an intervention that combines opioid overdose prevention, education and intervention that includes take home naloxone with brief behavioral change counseling. The study will recruit both heroin users (n=500) and pharmaceutical opioid users at elevated risk for overdose (n=500). Outcomes of interest include subsequent opioid overdoses and overdose risk behaviors.

Primary Aims

The primary aims are to test whether those who receive the intervention compared to standard care have: 1) Lower rates of opioid non-fatal and fatal overdose; 2) Reduce drug use, inappropriate medication use, and other overdose risk behaviors.

Secondary Aims

The secondary aims are to test whether those who receive the intervention compared to standard care have: 3) More appropriate health care utilization (e.g. fewer emergency department visits and admissions to inpatient care); 4) Lower total health care costs; 5) Determine the prevalence of HIV risk behaviors among heroin and pharmaceutical opioid users at risk for overdose and whether the intervention impacts these behaviors.

DETAILED DESCRIPTION:
Fatal overdoses involving pharmaceutical opioids have increased dramatically over the past decade, surpassing those related to heroin, and are the leading cause of drug overdose in much of the U.S. In Seattle-King County, 75% of drug overdoses involved pharmaceutical opioids and/or heroin in 2009. Opioid overdoses, heroin and pharmaceutical, are preventable and reversible. Research indicates that drug users and their partners can be successfully trained to recognize and reverse overdoses with naloxone (an opioid antagonist medicine or "antidote").

Despite active heroin overdose prevention, education and intervention programs with naloxone (OOPEN) in 15 states with thousands of overdose reversals and no serious adverse events, rigorous studies of these programs on rates of subsequent heroin overdoses have not been conducted. No OOPEN programs or studies have yet been implemented for pharmaceutical opioid users at elevated risk for overdose. The Emergency Department (ED) setting holds great promise for identifying and recruiting those at elevated risk of both heroin and pharmaceutical opioid overdose: 1) the ED study site for this proposal provides most services to those needing care for acute opioid related medical problems in Seattle, and 2) patients' need for urgent medical attention may heighten their concern about potential harms from opioids.

Unique to this setting is the potential to identify high risk pharmaceutical opioid users, a population that is difficult to locate and engage. ED interventions using brief behavior change counseling (BBCC) have been shown to significantly improve health behaviors such as alcohol use and injury, to increase entry into drug treatment as well as to reduce costs. Evidence is promising, but limited, regarding the impact of BBCC on opioid related risk behaviors.

This prospective, randomized ED trial will study the effectiveness of an intervention that combines OOPEN with BBCC for both heroin users (n=500) and pharmaceutical opioid users at elevated risk for overdose (n=500). The primary outcome is subsequent opioid overdoses, ascertained by follow up interviews conducted at 3, 6 and 12 months as well as via administrative records for up to 24 months (i.e. medical records, ambulance responses, and death certificates).

Primary Aims

The primary aims are to test whether those who receive the intervention compared to standard care have: 1) Lower rates of opioid non-fatal and fatal overdose; 2) Reduce drug use, inappropriate medication use, and other overdose risk behaviors.

Secondary Aims

The secondary aims are to test whether those who receive the intervention compared to standard care have: 3) More appropriate health care utilization (e.g. fewer emergency department visits and admissions to inpatient care); 4) Lower total health care costs; 5) Determine the prevalence of HIV risk behaviors among heroin and pharmaceutical opioid users at risk for overdose and whether the intervention impacts these behaviors.

ELIGIBILITY:
Inclusion Criteria:

Meets study definition of elevated risk of future opioid overdose

* Reason for visit is opioid overdose (regardless of frequency of use), or
* Use of pharmaceutical opioids not prescribed to the patient 2 or more times in the prior month, or
* Use of other opioids, alcohol, benzodiazepines or stimulants within two hours of using opioids 2 or more times in the prior month, or
* Average daily dose of prescribed opioids consumed is greater than10 mg morphine equivalent analgesic dose or higher for 15 or more days in the last 30.
* Enrolled in opioid substitution program (e.g. methadone or suboxone) and receiving doses.
* Use of heroin through any route of administration at least 2 times in the last 30 days (or if institutionalized recently, in the most recent month they were not institutionalized) with or without other risks being present.
* Use of pharmaceutical opioids at least 2 times in the last 30 days (or if institutionalized recently, in the most recent month they were not institutionalized) with other risks being present.
* Average daily dose of prescribed opioids consumed is 30 mg morphine equivalent analgesic dose or higher without other risks being present.(For adult medicine clinic patients only.)

Exclusion Criteria:

* Unwilling to allow further access to medical or drug treatment records.
* Inability to communicate in English.
* Current active suicidal ideation.
* Significant cognitive or psychiatric impairment (per judgment of clinical staff)
* Inability to provide adequate contact information to assist with follow-up.
* Under age 18 or over age 70 at time of recruitment.
* Not currently living in Washington State or planning to move from Washington State within the following year.
* Receiving treatment for sexual assault.
* Have non-expired take-home naloxone at home, on their person, or in their possessions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Harborview Medical Center, Seattle, Washington
  - Evergreen Treatment Services, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Banta-Green CJ, Coffin PO, Merrill JO, Sears JM, Dunn C, Floyd AS, Whiteside LK, Yanez ND, Donovan DM. Impacts of an opioid overdose prevention intervention delivered subsequent to acute care. Inj Prev. 2019 Jun;25(3):191-198. doi: 10.1136/injuryprev-2017-042676. Epub 2018 Feb 7. PMID 29436397

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention (OOPEN+BBCC) | Control
Started | 125 | 131
Completed | 115 | 126
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (OOPEN+BBCC) | Control | Total
Number analyzed (Participants) | 115 | 126 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.5) | 42.3 (11.5) | 41.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 69
  Male | 83 | 89 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 21 | 35
  Not Hispanic or Latino | 101 | 105 | 206
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 12
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 17 | 14 | 31
  White | 60 | 67 | 127
  More than one race | 18 | 19 | 37
  Unknown or Not Reported | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  United States | 115 | 126 | 241
Opioid overdose past 3 months [Count of Participants; unit: Participants] | 19 | 27 | 46

OUTCOME MEASURES:

1. Primary Outcome: Rate of Fatal Opioid Overdose
Description: Rate of fatal opioid overdose
Time Frame: One year
Population: Number of participants experiencing fatal opioid overdose.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 115 | 126
Participants | 2 | 6

2. Primary Outcome: Rate of Non-fatal Opioid Overdose
Description: Rate of non-fatal opioid overdose
Time Frame: One year
Population: Number of participants experiencing non-fatal opioid overdose.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 115 | 126
Participants | 22 | 27

3. Primary Outcome: Elapsed Time Until Opioid Overdose
Description: Elapsed time until opioid overdose
Time Frame: Up to1064 days
Population: Mean days to first overdose event
Measure: Mean (Full Range); unit: days
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 115 | 126
days | 870 [272 to 1064] | 836 [272 to 1064]

4. Primary Outcome: Change in Overdose Risk (Change in Opioid Use - Heroin)
Description: Determine whether changes in behavior occur that increase or decrease risk of future overdose. Behaviors being measured include the amount of opioids taken, the use of opioids alone, use of opioids with alcohol or other drugs or medications, possessing naloxone, use of opioids in an environment that supports continued opioid use.(Data table includes proportions at 3 month follow-up.)
Time Frame: 3 months
Population: Participants reporting change in heroin use: "Compared to the last time you spoke with research staff 3 months ago, do you use heroin..."
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 30 | 29
Participants
  More | 6 | 4
  Less | 14 | 17
  Same Amount | 7 | 7
  Don't Know | 3 | 1
  N/A (was not using previously) | 0 | 0

5. Primary Outcome: Change in Overdose Risk (Change in Opioid Use - Prescription-Type Opioids)
Description: as for outcome 4
Time Frame: 3 months
Population: Participants reporting change in prescription-type opioid use: "Compared to the last time you spoke with research staff 3 months ago, do you use prescription-type medications..."
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 35 | 39
Participants
  More | 7 | 9
  Less | 12 | 11
  Same Amount | 12 | 16
  Don't know Don't Know | 2 | 3
  N/A (was not using previously) | 2 | 0

6. Primary Outcome: Change in Overdose Risk (Using Alone When Taking Opioids)
Description: Determine whether changes in behavior occur that increase or decrease risk of future overdose. Behaviors being measured include the amount of opioids taken, the use of opioids alone, use of opioids with alcohol or other drugs or medications, possessing naloxone, use of opioids in an environment that supports continued opioid use. (Data table includes means at 3 month follow-up.)
Time Frame: 3 months
Population: Mean days using opioids alone, among people who used one or more days in the past 30, "In the past 30 days, how many days have you used opioids when nobody else was around?"
Measure: Mean (Standard Deviation); unit: days in the past 30
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 97 | 103
days in the past 30
  Baseline | 17.9 (10.5) | 15.6 (10.9)
  Follow-up: number analyzed (Participants) | 17 | 25
  Follow-up | 16.5 (10.9) | 16.7 (10.7)

7. Primary Outcome: Change in Overdose Risk (Use of Sedatives When Taking Opioids)
Description: Determine whether changes in behavior occur that increase or decrease risk of future overdose. Behaviors being measured include the amount of opioids taken, the use of opioids alone, use of opioids with alcohol or other drugs or medications, possessing naloxone, use of opioids in an environment that supports continued opioid use. (Data table includes proportions at 3 month follow-up.)
Time Frame: 3 months
Population: Use of sedatives when taking opioids, "When you use opioids, how often do you use sedatives or downers within 2 hours before or after?"
  .
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 125 | 131
Participants
  Baseline: Always | 11 | 11
  Baseline: Sometimes | 41 | 53
  Baseline: Never | 73 | 67
  Follow-up: Always: number analyzed (Participants) | 56 | 58
  Follow-up: Always | 2 | 2
  Follow-up: Sometimes: number analyzed (Participants) | 56 | 58
  Follow-up: Sometimes | 15 | 11
  Follow-up: Never: number analyzed (Participants) | 56 | 58
  Follow-up: Never | 39 | 45

8. Primary Outcome: Change in Overdose Risk (Use of Alcohol When Taking Opioids)
Description: as for outcome 4
Time Frame: 3 months
Population: Use of alcohol when taking opioids, "When you use opioids, how often do drink alcohol with 2 hours before or after?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 125 | 131
Participants
  Baseline: Always | 8 | 19
  Baseline: Sometimes | 31 | 35
  Baseline: Never | 86 | 77
  Follow-up: Always: number analyzed (Participants) | 57 | 58
  Follow-up: Always | 5 | 4
  Follow-up: Sometimes: number analyzed (Participants) | 57 | 58
  Follow-up: Sometimes | 9 | 9
  Follow-up: Never: number analyzed (Participants) | 57 | 58
  Follow-up: Never | 43 | 45

9. Secondary Outcome: Health Care Utilization (ED and Inpatient Admissions)
Description: Appropriate health care utilization (e.g. fewer emergency department visits and admissions to inpatient care)
Time Frame: One year (annual rate)
Population: Annual mean number per person
Measure: Mean (95% Confidence Interval); unit: annual visits
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 115 | 126
annual visits
  Emergency department visits | 4.96 [4.04 to 6.10] | 4.85 [3.96 to 5.93]
  Inpatient admissions | 1.29 [0.95 to 1.76] | 1.05 [0.80 to 1.39]

10. Secondary Outcome: Change in HIV Risk Behaviors (Condom Use)
Description: Determine whether change occurs in the number of sexual risk behaviors (such as engaging in intercourse without a condom) and/or injection use behaviors (such as sharing syringes) that may increase the risk of contracting HIV.(Data table includes proportions at 3 month follow-up.)
Time Frame: 3 months
Population: Frequency of condom use in the past 3 months, "In the past three months, how often did you use condoms when you had sex?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 71 | 73
Participants
  Baseline: All the time | 20 | 14
  Baseline: Most of the time | 8 | 6
  Baseline: Some of the time | 8 | 5
  Baseline: None of the time | 33 | 45
  Baseline: Not applicable/No sex past 3 months | 2 | 3
  Follow-up: number analyzed (Participants) | 29 | 25
  Follow-up: All the time | 12 | 5
  Follow-up: Most of the time | 0 | 1
  Follow-up: Some of the time | 3 | 1
  Follow-up: None of the time | 13 | 15
  Follow-up: Not applicable/No sex past 3 months | 1 | 3

11. Secondary Outcome: Change in HIV Risk Behaviors (Shared Syringes)
Description: Determine whether change occurs in the number of sexual risk behaviors (such as engaging in intercourse without a condom) and/or injection use behaviors (such as sharing syringes) that may increase the risk of contracting HIV. (Data table includes proportions at 3 month follow-up.)
Time Frame: 3 months
Population: Number of participants who shared syringes or injection supplies, "In the past three months, have you shared needles or works?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 102 | 97
Participants
  Baseline | 29 | 29
  Follow-up: number analyzed (Participants) | 37 | 32
  Follow-up | 11 | 4

12. Secondary Outcome: Change in Overdose Risk Behaviors and Perceptions (Take Home Naloxone)
Description: Change in overdose response including naloxone availability and change in overdose risk perceptions. (Data table includes proportions at 3 month follow-up.)
Time Frame: 3 Months
Population: Number of people with naloxone in the past 3 months, "At any time in the past 3 months did you have take-home naloxone?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 57 | 58
Participants | 41 | 10

13. Secondary Outcome: Change in Overdose Risk Behaviors and Perceptions (Likelihood of Overdose)
Description: as for outcome 12
Time Frame: 3 Months
Population: Perception of likelihood of opioid overdose, "How likely is it that you will experience an opiate overdose in the next year?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 64 | 63
Participants
  Baseline: Extremely/somewhat likely | 12 | 15
  Baseline: Not sure | 14 | 19
  Baseline: Extreme/somewhat unlikely | 38 | 29
  Follow-up: number analyzed (Participants) | 35 | 29
  Follow-up: Extremely/somewhat likely | 1 | 3
  Follow-up: Not sure | 17 | 6
  Follow-up: Extreme/somewhat unlikely | 17 | 20

14. Secondary Outcome: Change in Overdose Risk Behaviors and Perceptions (Concerned About Overdose)
Description: as for outcome 12
Time Frame: 3 Months
Population: Perception of concern about opioid overdose, "How concerned are you about YOU experiencing an overdose?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 64 | 63
Participants
  Baseline: Extremely/somewhat concerned | 24 | 28
  Baseline: Not sure | 1 | 3
  Baseline: Not very/at all concerned | 39 | 32
  Follow-up: number analyzed (Participants) | 35 | 29
  Follow-up: Extremely/somewhat concerned | 9 | 7
  Follow-up: Not sure | 2 | 0
  Follow-up: Not very/at all concerned | 24 | 22

15. Secondary Outcome: Subgroup Analyses - Change in HIV Risk Behaviors (Condom Use)
Description: Sub-group analyses- primary and secondary outcomes will be examined by homelessness status at baseline.(Data table includes proportions at 3 month follow-up.)
Time Frame: 3 months
Population: Frequency of condom use in the past 3 months by housing status. "In the past three months, how often did you use condoms when you had sex?"
Measure: Count of Participants; unit: Participants
Groups:
- Intervention (OOPEN+BBCC) - Permanent or Stable Housing; Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused: Study intervention, overdose prevention, education, intervention, brief behavioral change counseling, take-home naloxone, referral to local available resources.
  OOPEN+BBCC: Take-home naloxone is offered as part of a behavioral prevention intervention to reduce the occurrence of future opioid overdose.
- Control - Permanent or Stable Housing; Control - Temporary or Unstable Housing or Unhoused.: Standard of care, referral to local available resources.
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 10 | 19 | 12 | 13
Participants
  All the time | 4 | 8 | 2 | 3
  Most of the time | 0 | 0 | 0 | 1
  Some of the time | 1 | 2 | 1 | 0
  None of the time | 5 | 8 | 8 | 7
  Not applicable/No sex past 3 months | 0 | 1 | 1 | 2

16. Secondary Outcome: Subgroup Analyses - Change in HIV Risk Behaviors (Shared Syringes)
Description: as for outcome 15
Time Frame: 3 months
Population: Number of participants who shared syringes or injection supplies by housing status. "In the past three months, have you shared needles or works?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 11 | 26 | 15 | 17
Participants | 4 | 7 | 2 | 2

17. Secondary Outcome: Sub-group Analyses - Change in Overdose Risk (Change in Opioid Use - Heroin)
Description: as for outcome 15
Time Frame: 3 months
Population: Participants reporting change in heroin use by housing status: "Compared to the last time you spoke with research staff 3 months ago, do you use heroin..."
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 8 | 22 | 12 | 17
Participants
  More | 1 | 5 | 3 | 1
  Less | 4 | 10 | 6 | 11
  Same Amount | 2 | 5 | 3 | 4
  Don't Know | 1 | 2 | 0 | 1
  N/A (was not using previously) | 0 | 0 | 0 | 0

18. Secondary Outcome: Sub-group Analyses - Change in Overdose Risk (Change in Opioid Use - Prescription Type Opioids)
Description: as for outcome 15
Time Frame: 3 months
Population: Participants reporting change in prescription-type opioids by use by housing status: "Compared to the last time you spoke with research staff 3 months ago, do you use prescription type opioids..."
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 11 | 24 | 24 | 15
Participants
  More | 2 | 5 | 6 | 3
  Less | 3 | 9 | 7 | 4
  Same Amount | 5 | 7 | 10 | 6
  Don't Know | 1 | 1 | 1 | 2
  N/A (was not using previously) | 0 | 2 | 0 | 0

19. Secondary Outcome: Sub-group Analyses - Change in Overdose Risk (Using Alone When Taking Opioids)
Description: Sub-group analyses- primary and secondary outcomes will be examined by homelessness status at baseline.(Data table includes means at 3 month follow-up.)
Time Frame: 3 months
Population: Mean days using opioids alone, among people who used one or more days in the past 30 by housing status. "In the past 30 days, how many days have you used opioids when nobody else was around?"
Measure: Mean (Standard Deviation); unit: days in the past 30
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing | Control - Temporary or Unstable Housing or Unhoused
Number analyzed (Participants) | 8 | 9 | 14 | 11
days in the past 30 | 19.1 (10.8) | 14.2 (11.1) | 17.7 (10.8) | 15.4 (11.0)

20. Secondary Outcome: Subgroup Analyses- Change in Overdose Risk (Use of Sedatives When Taking Opioids)
Description: as for outcome 15
Time Frame: 3 months
Population: Use of sedatives when taking opioids by housing status. "When you use opioids, how often do you take sedatives or downers with 2 hours before or after?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 18 | 38 | 32 | 26
Participants
  Always | 1 | 1 | 0 | 2
  Sometimes | 6 | 9 | 3 | 8
  Never | 11 | 28 | 29 | 16

21. Secondary Outcome: Subgroup Analyses- Change in Overdose Risk (Use of Alcohol When Taking Opioids)
Description: as for outcome 15
Time Frame: 3 months
Population: Use of alcohol when taking opioids by housing status "When you use opioids, how often do drink alcohol with 2 hours before or after?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 18 | 39 | 32 | 26
Participants
  Always | 1 | 4 | 3 | 1
  Sometimes | 1 | 8 | 3 | 6
  Never | 16 | 27 | 26 | 19

22. Secondary Outcome: Sub-group Analyses - Change in Overdose Risk Behaviors and Perceptions (Take Home Naloxone)
Description: as for outcome 15
Time Frame: 3 Months
Population: Number of people with naloxone in the past 3 months by housing status. "At any time in the past 3 months did you have take-home naloxone?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 18 | 39 | 32 | 26
Participants | 11 | 30 | 4 | 6

23. Secondary Outcome: Sub-group Analyses- Change in Overdose Risk Behaviors and Perceptions (Likelihood of Overdose)
Description: as for outcome 15
Time Frame: 3 Months
Population: Perception of likelihood of opioid overdose by housing status. "How likely is it that you will experience an opiate overdose in the next year?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 8 | 27 | 16 | 13
Participants
  Extremely likely | 0 | 1 | 0 | 0
  Somewhat likely | 0 | 0 | 2 | 1
  Not sure | 2 | 5 | 3 | 3
  Somewhat unlikely | 3 | 7 | 3 | 1
  Extremely unlikely | 3 | 14 | 8 | 8

24. Secondary Outcome: Sub-group Analyses- Change in Overdose Risk Behaviors and Perceptions (Concerned About Overdose)
Description: as for outcome 15
Time Frame: 3 Months
Population: Perception of concern about opioid overdose by housing status. "How concerned are you about YOU experiencing an overdose?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (OOPEN+BBCC) - Permanent or Stable Housing | Intervention (OOPEN+BBCC) - Temporary or Unstable Housing or Unhoused | Control - Permanent or Stable Housing. | Control - Temporary or Unstable Housing or Unhoused.
Number analyzed (Participants) | 8 | 27 | 16 | 13
Participants
  Extremely concerned | 1 | 5 | 2 | 1
  Somewhat concerned | 1 | 2 | 3 | 1
  Not sure | 1 | 1 | 0 | 0
  Not very concerned | 4 | 6 | 4 | 2
  Not concerned at all | 1 | 13 | 7 | 9

25. Secondary Outcome: Health Care Costs
Description: Total health care costs
Time Frame: Two years
Population: Health care cost data were not obtained, therefore these analyses could not be conducted.
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Health Care Utilization
Description: Rate and elapsed time until initiation of buprenorphine or methadone maintenance. (for those not on treatment medications)
Time Frame: Two years
Population: Data for initiation of buprenorphine and methadone for those not on treatment medications were not obtained, therefore these analyses could not be conducted.
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Health Care Utilization
Description: Retention time on buprenorphine or methadone (for those on medications at baseline)
Time Frame: Two years
Population: Retention data for buprenorphine and methadone were not obtained, therefore these analyses could not be conducted.
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Opioid Overdose - Crossover Analysis
Description: Crossover analysis- Comparison group participants who obtain naloxone during the follow up period will be analyzed with those in the intervention arm and compared with those who did not obtain naloxone in the comparison arm to examine differences in overdose rates and elapsed time to overdose.
Time Frame: Two years
Population: Specific dates when naloxone was obtained were not collected, therefore these analyses could not be conducted.
Arm/Group | Intervention (OOPEN+BBCC) | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Three years.
Description: In this study, potential adverse events that may be related to the study would be an increase in emotional distress in relation to discussion of past or current drug use behaviors or side effects of naloxone.
Arm/Group | Intervention (OOPEN+BBCC) | Control
All-Cause Mortality (participants affected / at risk) | 10/115 | 13/126
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/126
Other Adverse Events (participants affected / at risk) | 0/115 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT01788306/Prot_SAP_000.pdf